CLINICAL TRIAL: NCT02373176
Title: [14C] PRC-4016 (Icosabutate) - A Phase I, Open-label Study of the Absorption, Metabolism and Excretion Following Oral Dosing to Healthy Male Subjects.
Brief Title: [14C] Icosabutate -A Phase I Absorption, Metabolism and Excretion Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pronova BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CTN401614102
Record Dates: First submitted 2015-02-09; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
MeSH Terms: interventions — icosabutate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C] PRC-4016 (Icosabutate) (Experimental): Investigational medicinal product (IMP), [14C] PRC-4016 (Icosabutate) solution (600 mg in 2 mL, 200.0 μCi [7.4 MBq]). The radiochemical purity of [14C]PRC-4016 will be at least 97%.
  Interventions: Drug: [14C]PRC 4016 (Icosabutate)

INTERVENTIONS:
Drug: [14C]PRC 4016 (Icosabutate) — Single oral dose
  Other Names: Icosabutate

SUMMARY:
[14C]PRC-4016 (Icosabutate) - A Phase I, Open-Label Study of the Absorption, Metabolism and Excretion Following Oral Dosing to Healthy Male Subjects.

Objective: To evaluate the pharmacokinetics of total radioactivity in blood and plasma and PRB-01022 (icosabutate) (unchanged drug) in plasma following a single oral administration of [14C]PRC-4016 to healthy male subjects.

To obtain a mass balance of oral [14C]PRC-4016 by quantifying the urinary and faecal excretion of radioactivity.

To examine the profile of metabolites in plasma, urine and faeces. To further assess the safety and tolerability of a single oral dose of [14C]PRC 4016 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* males
* any ethnic origin
* age 35-60
* BMI 18-35 kg/m2
* generally in good health
* signed informed consent

Exclusion Criteria:

* subjects or subjects partners not willing to use appropriate contraception
* subjects who have received prescribed systemic or topical medication within 14 days of dosing
* subjects who have used non-prescribed systemic or topical medication within 7 days of dosing
* subjects who have received any medication incl. St. Johns Worth within 30 days of dose administration.
* subjects participating in clinical trial currently or within past 3 months.
* recent blood donation
* history of drug allergy or clinically significant allergic disease
* BP and pulse outside reference range
* high consumption of alcohol
* high consumption og tobacco
* clinically significant disorder or clinically significant disease within 4 weeks of dosing.
* serum hepatitis, HIV or abnormal ECG
* subjects exposed to radiation as a result of their occupation
* subjects who have received radiolabelled material within 12 months
* subjects earlier taken part in the study or withdrawn from study ot not suitable for enrolment according to investigator.

Ages: 35 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area under curve for total 14C labelled PRC-4016 in whole blood and plasma. | Up to 168 hours post-dose
  Blood sampling
Peak plasma concentration of 14C labelled PRC-4016 (icosabutate) | Up to 168 hours post-dose
  Blood sampling
Quantifying urinary and faecal excretion of 14C labelled PRC-4016 | Up to 168 hours post-dose
  Urine- and faecal collection

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of a single dose oral 14C PRC-4016 (icosabutate) | During entire study, screening till Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MD PhD, Principal Investigator — Covance Clinical research Unit
Locations (1):
- Covance Clinical research Unit (CRU) Ltd,Springfield House, Hyde street, Leeds, United Kingdom